CLINICAL TRIAL: NCT04422587
Title: Evaluation of the COVID-19 Infection Response in Patients Admitted to the Emergency Department for Dyspnea
Acronym: EPRICOD
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0149
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Emergencies
Keywords: COVID-19; diagnostic strategy; acute dyspnea
MeSH Terms: conditions — Emergencies; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RECOP unit patient: All patients admit in RECOP unit for dyspnea can be included in this study if patient is agree. Then, doctor collects demographic variables, the usual history and treatments, the characteristics of the episode (symptomatology, evolution, treatment taken) and the data from the initial clinical examination will be identified.
  Interventions: Other: RECOP unit patient

INTERVENTIONS:
Other: RECOP unit patient — All patients admit in RECOP unit for dyspnea can be included in this study if patient is agree. Then, doctor collects demographic variables, the usual history and treatments, the characteristics of the episode (symptomatology, evolution, treatment taken) and the data from the initial clinical examination will be identified.

SUMMARY:
This research aims to improve our knowledge of the epidemiology of patients consulting in the COvid-19 Possible REspiratory Units (RECOP unit). Indeed, the epidemic linked to COVID-19 affects France and impacts its health system. The reception of all intermediate patients will be on the Emergency Structures (SU). Indeed, the French healthcare system centralizes unscheduled urgent care on the ER. The aspecific respiratory symptomatology in "intermediate" patients indicates them all the more at an admission to SU or the diagnostic approach to respiratory difficulty may be carried out.

A central issue of this diagnostic strategy will be to be rapid, since the diagnosis will have to be made in the context of significant flows, with a need to quickly refer patients to the most suitable downstream service, while limiting the risk contamination of caregivers and vulnerable patients if a COVID-19 + patient is admitted to an unsuitable service. However, virological tests do not currently allow rapid results for COVID-19.

Research project of investigatory aims to develop a predictive model of the risk of being COVID-19 positive for patients admitted to the emergency room for acute dyspnea.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 15 years admitted to the RECOP unit for dyspnea

Exclusion Criteria:

* Patient admitted to shock for respiratory distress requiring immediate respiratory support.
* Patient under justice safeguard

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patient admitted to the RECOP unit for dyspnea will be inclued in this clinical trial
Sampling Method: Non-Probability Sample
Enrollment: 1860 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-07 (Actual)

PRIMARY OUTCOMES:
Develop a predictive model of the risk of being COVID-19 for patients admitted to the emergency room for dyspnea | inclusion day
  demographic variables, usual history and treatments, episode characteristics (symptomatology, evolution, treatment taken) and data from the initial clinical examination will be collected by doctor

SECONDARY OUTCOMES:
Describe the characteristics of patients admitted to reCOP units according to their virological status | 30 days
  The COVID-19 virological condition will be taken with PCR tests on naso-pharyngeal samples or on sputum for patients taking
Virological status | 30 days
  Virological status will be collected by a phone call at the patient
Mortality status | 30 days
  Mortality status will be collected by a phone call at the patient

CONTACTS AND LOCATIONS:
Overall Officials: Paul-Henri Auboiroux, MD, Principal Investigator — University Hospital of Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No